CLINICAL TRIAL: NCT05749653
Title: Impact of a Bi-annual Community-directed Treatment With Ivermectin Programme on the Incidence of Epilepsy in an Onchocerciasis-endemic Area of Mahenge, Tanzania: a Population-based Prospective Study
Brief Title: Impact of a Bi-annual CDTI on the Incidence of Epilepsy in an Onchocerciasis-endemic Area
Acronym: OAETanzania
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiteit Antwerpen (Other)
Responsible Party: Principal Investigator, Robert Colebunders, Emeritus professor, head NSETHIO research group, Global Health institute, Universiteit Antwerpen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: B300201837863
Record Dates: First submitted 2023-02-17; First posted 2023-03-01 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Onchocerciasis; Epilepsy
MeSH Terms: conditions — Onchocerciasis; Epilepsy

STUDY DESIGN:
Intervention Model Description: population based study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- bi-annual CDTI (Other): bi-annual CDTI with high coverage
  Interventions: Drug: Bi-annual CDTI

INTERVENTIONS:
Drug: Bi-annual CDTI — Bi-annual CDTI

SUMMARY:
Onchocerciasis is a neglected tropical disease associated with epilepsy, particularly in areas of high Onchocerciasis volvulus transmission. Onchocerciasis-associated epilepsy is characterised by seizures that start between the ages of five to 18 years. The tropical disease can be controlled through community-directed treatment with ivermectin (CDTi). Mahenge, in Tanzania, had a high prevalence of onchocerciasis and epilepsy despite more than 20 years of annual CDTi. Hence, the Tanzanian Neglected Tropical Diseases Control Programme has switched from annual to bi-annually CDTi since 2019. After this switch, the CDTi coverage increased and was sustained in both ivermectin rounds in 2021, and the number of new epilepsy cases decreased. The latter were persons who did not take ivermectin the year they had the first seizures. Hence, all ivermectin-eligible children at risk of onchocerciasis should take ivermectin at least annually. Overall, increasing the frequency and coverage of the CDTi programme should be considered in onchocerciasis-endemic areas with a high prevalence of epilepsy.

DETAILED DESCRIPTION:
Background: Community-directed treatment with ivermectin (CDTi) is used to eliminate onchocerciasis. However, despite 25 years of annual CDTi in Mahenge, Tanzania, the prevalence of onchocerciasis and onchocerciasis-associated epilepsy remained high in certain rural villages. Therefore, in 2019, bi-annual CDTi was introduced in the area. This study assessed the impact of the programme on the incidence of epilepsy in four villages.

Methodology: Door-to-door epilepsy surveys were conducted prior to (2017/18) and after (2021) implementing bi-annual CDTi. All household members were screened for epilepsy symptoms using a validated questionnaire, and suspected cases were examined by a medical doctor to confirm/reject the diagnosis of epilepsy. The prevalence and annual incidence of epilepsy, including nodding syndrome, were calculated with 95% Wilson confidence intervals with continuity correction. The latter was also done for CDTi coverage in 2021.

ELIGIBILITY:
Inclusion Criteria: whole population -

Exclusion Criteria: No

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 6500 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Epilepsy incidence | 3 years
  Number of new epilepsy cases per month

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Mmbando, PhD, Principal Investigator — National Institute of Medical Research, Tanga
Locations (1):
- National Institute of Medical Research, Tanga, Tanzania

IPD SHARING:
Plan to Share IPD: No
After de-identification (text, tables, figures, and appendices), all individual participant data underlying the results reported in this article will be made available immediately and indefinitely via the Zenodo repository following publication for anyone who wishes to access the data for any purpose.